CLINICAL TRIAL: NCT03103295
Title: Safety and Efficacy Study of Traumatic Bone Defects Treatment With Use of 3D Tissue Engineered Equivalent.
Brief Title: 3D Tissue Engineered Bone Equivalent for Treatment of Traumatic Bone Defects
Acronym: 3-D-TEBE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: A.A. Partners, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-P2-14
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Bone Defects
Keywords: tissue engineering,; regeneration,; repair,; traumatic bone defects,; regenerative therapy

STUDY DESIGN:
Masking Description: Open
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3D-Tissue Engineered Bone Equivalent (Experimental): Patients with bone defects of critical size of long bones
  3D Tissue Engineered Bone Equivalent: allogeneic or xenogeneic partially demineralized bone matrix (DBM) and plasma-derived fibrin gel seeded with autologous cultured bone marrow-derived multipotent mesenchymal stromal cells (BM-MSCs), periosteal progenitor cells (PPCs), peripheral blood-derived endothelial progenitor cells (PB-EPCs).
  Interventions: Biological: 3D-Tissue Engineered Bone Equivalent

INTERVENTIONS:
Biological: 3D-Tissue Engineered Bone Equivalent — Administrated for operative delivery of 3D-Tissue Engineered Bone Equivalent
  Other Names: Tissue-engineered bone-like construct transplantation

SUMMARY:
This study investigates safety and efficacy of traumatic bone defects treatment with use of 3D tissue engineered bone equivalent (3D-TEBE).

The aim of this study is to evaluate 3D-TEBE transplantation as a safe and efficient treatment for patients with traumatic long bone defects of critical size.

DETAILED DESCRIPTION:
This new method of critical sized long bone defects treatment is under clinical development. Treatment of critical sized bone defects is an actual clinical challenge. The "gold standard" in this case is autologous bone grafting. The method disadvantage is associated with limited donor bone resources. Based on our preliminary clinical trial positive results on use of autologous cultured bone marrow-derived multipotent mesenchymal stromal cells (BM-MSCs) in traumatology, our aim was to develop 3D tissue-engineered bone equivalent transplantation technology for restoration of critical sized bone defects. The proposed 3D-TEBE transplantation for bone defects of critical size treatment expecting to restore the bone integrity, form new bone tissue in a site of bone defect, and reduce the rehabilitation period of a patient.

The data obtained from this study will have practical implications for the treatment of reparative osteogenesis alterations and will be based on the principles of evidence-based medicine

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* Patients with long bone defects of critical size of the traumatic genesis;
* Lack of consolidation of bone fragments for at least 9 months;
* At least two attempts to achieve bone consolidation using traditional methods of treatment;
* A negative pregnancy test at women of childbearing age;
* Confirmation of participation in the study by signing The Written Informed Consent, personally or through a responsible caretaker;

Exclusion Criteria:

* The infection in the area of bone defect;
* History of prior cancer;
* Diabetes;
* Severe chronic liver diseases or kidneys disease in history
* Pregnancy;
* The presence of vascular, endocrine and somatic pathology which has a direct impact on the osteoreparation;
* Any other physical diseases in decompensation or subcompensation, or those that are rated as severe or moderate;
* Therapeutic issues or psychiatric disorders of a patient which would make the subject unsuitable to participate in this study or to complete it;
* Participation in another clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11-20 (Actual); Primary Completion 2018-12-20 (Estimated); Study Completion 2018-12-20 (Estimated)

PRIMARY OUTCOMES:
Radiographic and MRI assessment in progression | 12 months +3 years following 3D Tissue Engineered Bone Equivalent grafting
  Radiological and MRI progression of consolidation of bone fragments

SECONDARY OUTCOMES:
Reduction of pain using VAS | 6 months
  Patients feel less pain during use of fractured limb
Cost analysis based on length of hospital stay | 6 months
  Cost benefit of 3D-TEBE transplantation by reduction of hospital admission time

CONTACTS AND LOCATIONS:
Overall Officials: Volodymyr M. Oksymets, MD,PhD,DSci, Principal Investigator — LIMITED LIABILITY COMPANY "A.A. PARTNERS" (Medical company ilaya® ),
Locations (1):
- LIMITED LIABILITY COMPANY "A.A. PARTNERS" (Medical company ilaya®), Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Volodymyr Oksymets, Dmytro Zubov, Roman Vasyliev, Anzhela Rodnichenko, Olga Gubar, Alena Zlatska, Vitaliy Oksymets. Tissue-engineered bone for traumatology and orthopedics: biotechnology aspects and clinical outcomes.//Absract book. Posters. 37th SICOT — http://artsloi.sicot.org/rome/Abstract-Book-Posters.pdf